CLINICAL TRIAL: NCT03057431
Title: Randomized Double-blind Placebo-controlled Trial Assessing the Efficacy of Standard and Low Dose Hydrochlorothiazide Treatment in the Prevention of Recurrent Nephrolithiasis
Brief Title: Hydrochlorothiazide for Kidney Stone Recurrence Prevention
Acronym: NOSTONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-01475
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Nephrolithiasis
Keywords: kidney stones; hydrochlorothiazide
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi | interventions — Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Once daily for 3 years
  Interventions: Drug: Placebo oral capsule
- 12.5 mg hydrochlorothiazide (Experimental): Once daily for 3 years
  Interventions: Drug: 12.5 mg hydrochlorothiazide
- 25.0 mg hydrochlorothiazide (Experimental): Once daily for 3 years
  Interventions: Drug: 25.0 mg hydrochlorothiazide
- 50.0 mg hydrochlorothiazide (Experimental): Once daily for 3 years
  Interventions: Drug: 50.0 mg hydrochlorothiazide

INTERVENTIONS:
Drug: Placebo oral capsule — Once daily for 3 years
  Arms: Placebo
Drug: 12.5 mg hydrochlorothiazide — Once daily for 3 years
  Arms: 12.5 mg hydrochlorothiazide
Drug: 25.0 mg hydrochlorothiazide — Once daily for 3 years
  Arms: 25.0 mg hydrochlorothiazide
Drug: 50.0 mg hydrochlorothiazide — Once daily for 3 years
  Arms: 50.0 mg hydrochlorothiazide

SUMMARY:
The investigators plan to assess the efficacy of standard and low dose HCTZ treatment in the recurrence prevention of calcium-containing kidney stones. More specifically, the investigators aim to assess the dose-response relationship for three different dosages of HCTZ.

Study intervention: HCTZ 12.5 mg, 25 mg or 50 mg once daily per os for 24 or 36 months. In addition, all patients in HCTZ treatment arms will receive state-of-the-art non-pharmacologic recommendations for stone prevention according to current guidelines.

Control intervention: Placebo once daily per os for 24 to 36 months. In addition, all patients in the placebo arm will receive state-of-the-art non-pharmacologic recommendations for stone prevention according to current guidelines.

DETAILED DESCRIPTION:
Nephrolithiasis is a global healthcare problem with a current lifetime risk of 18.8% in men and 9.4% in women. Without specific treatment, 5- and 20-year recurrence rates are 40% and 75%, respectively. Given the high cost of medical treatments and surgical interventions as well as the morbidity related to symptomatic stone disease, medical prophylaxis for stone recurrence is an attractive approach.

About 80-90% of stones are composed of calcium oxalate with various admixtures of calcium phosphate. Increased excretion of calcium in the urine, hypercalciuria, is the most common metabolic abnormality encountered in patients with recurrent nephrolithiasis. Thiazide diuretics have been the cornerstone of pharmacologic metaphylaxis for more than 40 years. The effect of thiazides to reduce the risk of stone recurrence has been attributed to their ability to decrease urinary calcium excretion. However, other factors, such as reduction of urinary pH and urinary oxalate excretion, probably contribute to this effect. Efficacy of thiazides on recurrence prevention of calcareous nephrolithiasis was tested in 11 randomized controlled trials (RCTs). With the exception of two trials, thiazides significantly reduced stone recurrence. Most of these trials are from the 1980's and 90's and the cumulative number of patients studied is remarkably low for such a prevalent disease. Our systematic review of these RCTs revealed major methodological deficiencies in all trials, including: lack of double-blinding and intention-to-treat analysis, unclear allocation concealment, lack of adverse event and drop out reporting and unknown baseline risk of disease severity. Furthermore, high doses of thiazides were employed in all trials, in the case of the best studied thiazide, hydrochlorothiazide (HCTZ), up to 100 mg daily. At such high doses, side effects occur frequently. Nowadays, thiazides are widely used in the treatment of recurrent nephrolithiasis and arterial hypertension, but at significantly lower doses. In the case of recurrent nephrolithiasis, however, this practice is not supported by randomized evidence and consequently, the investigators do not know whether the currently employed low dose thiazide regimens are effective in reducing the risk for stone recurrence.

Thus, evidence for benefits and harms of thiazide diuretics in the prevention of calcium-containing kidney stones in general remains unclear. In addition, the efficacy of the currently employed low dose thiazide regimens to prevent stone recurrence is not known.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature
2. Age 18 years or older
3. Recurrent kidney stone disease (≥ 2 stone events within the last 10 years prior to randomization)
4. Any past kidney stone containing 50% or more of calcium oxalate, calcium phosphate or a mixture of both

Exclusion Criteria:

1. Pharmacologic prevention for stone recurrence less than 3 months prior to randomization
2. Patients with secondary causes of recurrent calcareous nephrolithiasis including:

   * Severe eating disorders (anorexia or bulimia)
   * Chronic inflammatory bowel disease, bariatric surgery, intestinal surgery with malabsorption or chronic diarrheal status
   * Sarcoidosis
   * Primary hyperparathyroidism
   * Complete distal tubular acidosis
   * Active malignancy
3. Patients with the following medications:

   * Thiazide or loop diuretics
   * Carbonic anhydrase inhibitors (including topiramate)
   * Xanthine oxidase inhibitors (febuxostat or allopurinol)
   * Alkali, including potassium citrate or sodium bicarbonate
   * Treatment with 1,25-OH Vitamin D (calcitriol)
   * Calcium supplementation
   * Bisphosphonates
   * Denosumab
   * Teriparatide
   * Glucocorticoids
4. Obstructive uropathy, if not treated successfully
5. Urinary tract infection, if not treated successfully
6. Chronic kidney disease (defined as CKD-EPI eGFR < 30 mL/min per 1,73 m2 body surface area for more than 3 months)
7. Patients with a kidney transplant
8. > 3 gout arthritis episodes within one year prior to randomisation or gout arthritis requiring uric acid lowering therapy
9. Cystinuria at screening
10. Hypokalemia (blood potassium level < 3 mmol/L) at screening
11. Hyponatremia (blood sodium level < 125 mmol/L) at screening
12. Pregnant and lactating women [pregnancy test to be performed for women of child-bearing potential (defined as women who are not surgically sterilized/ hysterectomized, and/ or who are postmenopausal for less than 12 months)]
13. Previous (within 3 months prior to randomization) or concomitant participation in another interventional clinical trial
14. Inability to understand and follow the protocol
15. Known allergy to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fuster, Prof MD, Principal Investigator — Division of Nephrology and Hypertension, Bern University Hospital, Bern, Switzerland
Locations (12):
- Switzerland (12):
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel
  - Ospedale Regionale di Bellinzona e Valli (San Giovanni), Bellinzona
  - Bern University Hospital (Inselspital), Bern
  - Kantonsspital Graubünden, Chur
  - Hôpitaux universitaires de Genève (HUG), Geneva
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Ospedale Regionale di Lugano (Civico), Lugano
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hôpital de Sion, Sion
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhayat NA, Bonny O, Roth B, Christe A, Ritter A, Mohebbi N, Faller N, Pellegrini L, Bedino G, Venzin RM, Grosse P, Husler C, Koneth I, Bucher C, Del Giorno R, Gabutti L, Mayr M, Odermatt U, Buchkremer F, Ernandez T, Stoermann-Chopard C, Teta D, Vogt B, Roumet M, Tamo L, Cereghetti GM, Trelle S, Fuster DG. Hydrochlorothiazide and Prevention of Kidney-Stone Recurrence. N Engl J Med. 2023 Mar 2;388(9):781-791. doi: 10.1056/NEJMoa2209275. PMID 36856614
- [Derived] Stritt K, Fuster DG, Dhayat NA, Bonny O, Faller N, Christe A, Taha A, Ochs V, Ortlieb N, Roth B; on behalf of the NOSTONE Study. Risk Factors of Asymptomatic Kidney Stone Passage in Adults with Recurrent Kidney Stones. Clin J Am Soc Nephrol. 2024 Sep 1;19(9):1130-1137. doi: 10.2215/CJN.0000000000000496. Epub 2024 Jul 19. PMID 39028573
- [Derived] Dhayat NA, Faller N, Bonny O, Mohebbi N, Ritter A, Pellegrini L, Bedino G, Schonholzer C, Venzin RM, Husler C, Koneth I, Del Giorno R, Gabutti L, Amico P, Mayr M, Odermatt U, Buchkremer F, Ernandez T, Stoermann-Chopard C, Teta D, Rintelen F, Roumet M, Irincheeva I, Trelle S, Tamo L, Roth B, Vogt B, Fuster DG. Efficacy of standard and low dose hydrochlorothiazide in the recurrence prevention of calcium nephrolithiasis (NOSTONE trial): protocol for a randomized double-blind placebo-controlled trial. BMC Nephrol. 2018 Dec 10;19(1):349. doi: 10.1186/s12882-018-1144-6. PMID 30526528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Specified in the protocol
Pre-assignment Details: No significant events.
Period: Overall Study
Arm/Group | Placebo | 12.5 mg Hydrochlorothiazide | 25.0 mg Hydrochlorothiazide | 50.0 mg Hydrochlorothiazide
Started | 102 | 105 | 108 | 101
Completed | 95 | 102 | 104 | 92
Not Completed | 7 | 3 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 12.5 mg Hydrochlorothiazide | 25.0 mg Hydrochlorothiazide | 50.0 mg Hydrochlorothiazide | Total
Number analyzed (Participants) | 102 | 105 | 108 | 101 | 416
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [35 to 55] | 49 [40 to 57] | 48 [39 to 56] | 50 [42 to 55] | 49 [39 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 16 | 22 | 21 | 85
  Male | 76 | 89 | 86 | 80 | 331
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 102 | 105 | 108 | 101 | 416
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 102 | 105 | 108 | 101 | 416

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stone Recurrences
Description: Composite of symptomatic or radiological recurrences, defined as either a symptomatic kidney stone passage or radiological kidney stone recurrence on CT.
  Symptomatic recurrence was defined as the visible passage of a stone with or without accompanying typical symptoms (such as flank or loin pain and hematuria) or as the presence of a symptomatic or asymptomatic stone that was determined to require surgical removal. If a patient had symptoms during the trial that were suggestive of a possible stone passage but no visible stone had been observed, local investigators evaluated the symptoms of the patient and judged whether a stone passage had occurred. Radiological recurrence was defined as a new stone formed or enlargement of a preexisting stone.
Time Frame: After 3 years
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 12.5 mg Hydrochlorothiazide | 25.0 mg Hydrochlorothiazide | 50.0 mg Hydrochlorothiazide
Number analyzed (Participants) | 102 | 105 | 108 | 101
Participants | 60 | 62 | 61 | 49

2. Secondary Outcome: Number of Symptomatic Stone Recurrences
Description: Symptomatic recurrence was defined as the visible passage of a stone with or without accompanying typical symptoms (such as flank or loin pain and hematuria) or as the presence of a symptomatic or asymptomatic stone that was determined to require surgical removal. If a patient had symptoms during the trial that were suggestive of a possible stone passage but no visible stone had been observed, local investigators evaluated the symptoms of the patient and judged whether a stone passage had occurred.
Time Frame: After 3 years
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 12.5 mg Hydrochlorothiazide | 25.0 mg Hydrochlorothiazide | 50.0 mg Hydrochlorothiazide
Number analyzed (Participants) | 102 | 105 | 108 | 101
Participants | 35 | 40 | 43 | 28

3. Secondary Outcome: Number of Radiologic Stone Recurrences.
Description: Radiological stone recurrence was defined as a new stone formed or enlargement of a preexisting stone (assessed by low-dose CT of the kidney at the end of the study compared to the low-dose CT of the kidney at the baseline visit).
Time Frame: After 3 years
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 12.5 mg Hydrochlorothiazide | 25.0 mg Hydrochlorothiazide | 50.0 mg Hydrochlorothiazide
Number analyzed (Participants) | 102 | 105 | 108 | 101
Participants | 46 | 44 | 32 | 31

ADVERSE EVENTS:
Time Frame: Every 3 months until study end at 3 years.
Description: We used standard definitions.
Arm/Group | Placebo | 12.5 mg Hydrochlorothiazide | 25.0 mg Hydrochlorothiazide | 50.0 mg Hydrochlorothiazide
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/105 | 0/108 | 0/101
Serious Adverse Events (participants affected / at risk) | 2/102 | 0/105 | 2/108 | 1/101
Other Adverse Events (participants affected / at risk) | 1/102 | 2/105 | 7/108 | 2/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | 12.5 mg Hydrochlorothiazide (N=105) | 25.0 mg Hydrochlorothiazide (N=108) | 50.0 mg Hydrochlorothiazide (N=101)
Pregnancy (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | 12.5 mg Hydrochlorothiazide (N=105) | 25.0 mg Hydrochlorothiazide (N=108) | 50.0 mg Hydrochlorothiazide (N=101)
New onset diabetes mellitus (Endocrine disorders) | 1 (1) | 2 (2) | 7 (7) | 2 (2)

LIMITATIONS AND CAVEATS:
Limited ethnic diversity, underrepresentation of women, trial duration of 3 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT03057431/Prot_SAP_000.pdf